CLINICAL TRIAL: NCT01604135
Title: Collagen Crosslinking for Keratoconus - a Randomized Controlled Clinical Trial
Acronym: CXL-RCT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Wolf K Wonneberger, MD, Ophthalmologist, Cornea and External Diseases Team, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNR-949-11
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Keratoconus
Keywords: Collagen crosslinking; Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corneal Collagen Crosslinking (Active Comparator): The keratokonic eye which progresses most is included and randomized. Significant progression is defined in the eligibility criteria section. If randomized to the treatment arm the cornea is treated with collagen crosslinking as described below.
  Interventions: Device: Corneal Collagen Crosslinking
- Control group (No Intervention): The keratokonic eye which progresses most is included and randomized to either the treatment group (CXL) or the control group.

INTERVENTIONS:
Device: Corneal Collagen Crosslinking — Keratoconic corneas that show significant progression as specified in the inclusion criteria section will receive one single treatment with CXL if randomized to the treatment arm. A treatment protocol based on 30 minutes dropping with riboflavin/dextran solution and 10 minutes UV-illumination treatment will be used.
  Other Names: Cross-Linking Procedure UV-X 2000; UV-X 2000 Illumination system; Innocross-R 0.1% dextran 20% solution; Innocross-R hypotonic riboflavin 0.1%
  Arms: Corneal Collagen Crosslinking

SUMMARY:
The purpose of this study is to determine whether corneal collagen crosslinking is effective in the treatment of progressive keratoconus.

DETAILED DESCRIPTION:
Keratoconus is a noninflammatory, asymmetrical, progressive corneal ectasia caused by biomechanical instability of the corneal stroma. Treatment modalities are primarily glasses or contact lenses. It has been estimated that one out of five patients will progress to such an extent that a corneal transplant is necessary to regain useful vision.

Corneal collagen crosslinking (CXL) is a treatment modality that intends to halt progression of keratoconus. This study investigates the efficacy av CXL in stabilizing the cornea in keratoconus by means of a randomized controlled clinical trial.

Participants are eligible for inclusion if progressive keratoconus is confirmed and the inclusion criteria are met. Follow-up after inclusion is at 1 week (treatment group), 1, 3, 6 and 12 months. Pre- and post-inclusion examinations include measurement of uncorrected distance visual acuity (UCDVA), best spectacle corrected distance visual acuity (BSCDVA), Scheimpflug-topography and slitlamp examination.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus diagnosis determined clinically and topographically (KISA%- index)
* Significant progression is defined as change (increase) of Kmax by at least

  1D from baseline at 6 months and/or change (increase) of Sim-K-ast by at least 1D from baseline at 6 months. Kmax is defined as the steepest radius of curvature (either the maximum simulated K-reading or the maximum K-reading in the 3-mm zone or the 5-mm zone) of the anterior corneal surface that progressed the most during 6 months observation
* Ability to stop contact lens (rigid and soft) wear at least two weeks prior to next exam
* Signed written informed consent

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Breast feeding
* History of corneal surgery
* History of ocular herpes simplex infection
* Minimal corneal thickness < 300 micrometers
* Recurrent corneal erosions
* Other corneal (e g endothelial) or conjunktival diseases
* Neurodermatitis
* Severe forms av atopic disease
* Collagenoses, autoimmune or other systemic disease
* Systemic treatment with high doses of steroids
* Severe scarring och striae of the cornea

Relative exclusion criteria:

* Kmax > 58D
* Minimal corneal thickness < 400 micrometers (a modified CXL-treatment will be used swelling the cornea before UV-illumination treatment).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Kmax | 12 months
  Kmax is defined as the steepest radius of curvature of the anterior corneal surface. It is measured by Scheimpflug-topography (Pentacam, Oculus Inc.). An increase of less than 1 diopter (D) from baseline at 12 months is defined as non-progression.

SECONDARY OUTCOMES:
Sim-K-astigmatism | 12 months
  Sim-K-astigmatism (Sim-K-ast) is defined as the absolute amount of anterior corneal astigmatism related to the Sim-Ks as measured by Scheimpflug-topography (Pentacam, Oculus Inc.). An increase of less than 1 D from baseline at 12 months is defined as non progression.
MRSE | 12 months
  Manifest Refractive Spherical Equivalent. The spherical equivalent is calculated by algebraic addition of the spherical power and half the cylindrical power of an eye. An eye with a specific spherical equivalent power has the closest overall effect to a given toric lens. A decrease of less than 0.5 D from baseline at 12 months is defined as non-progression.
UCDVA | 12 months
  UCDVA is defined as the uncorrected distance visual acuity measured with an Early Treatment of Diabetic Retinopathy Study (ETDRS)-chart and expressed in numbers of letters. A decrease of less than 5 letters (one line) from baseline at 12 months is defined as stable BCDVA.
BSCDVA | 12 months
  BSCDVA is defined as the the best spectacle corrected distance visual acuity measured with an ETDRS-chart and expressed in numbers of letters. A decrease of less than 5 letters (one line) from baseline at 12 months is defined as stable BCDVA.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Zetterberg, MD, PhD, Study Chair — Sahlgrenska University Hospital; Margareta Claesson, MD, PhD, Study Director — Sahlgrenska University Hospital
Locations (1):
- Department of Ophthalmology, Sahlgrenska University Hospital, Mölndal, Västra Götalandsregionen, Sweden

REFERENCES:
- [Background] Hersh PS, Greenstein SA, Fry KL. Corneal collagen crosslinking for keratoconus and corneal ectasia: One-year results. J Cataract Refract Surg. 2011 Jan;37(1):149-60. doi: 10.1016/j.jcrs.2010.07.030. PMID 21183110
- [Background] Greenstein SA, Fry KL, Hersh PS. Corneal topography indices after corneal collagen crosslinking for keratoconus and corneal ectasia: one-year results. J Cataract Refract Surg. 2011 Jul;37(7):1282-90. doi: 10.1016/j.jcrs.2011.01.029. PMID 21700105
- [Background] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Background] Wittig-Silva C, Chan E, Islam FM, Wu T, Whiting M, Snibson GR. A randomized, controlled trial of corneal collagen cross-linking in progressive keratoconus: three-year results. Ophthalmology. 2014 Apr;121(4):812-21. doi: 10.1016/j.ophtha.2013.10.028. Epub 2014 Jan 6. PMID 24393351